CLINICAL TRIAL: NCT01721746
Title: A Randomized Open-Label Phase 3 Trial of BMS-936558 (Nivolumab) Versus Investigator's Choice in Advanced (Unresectable or Metastatic) Melanoma Patients Progressing Post Anti-CTLA-4 Therapy
Brief Title: A Study to Compare BMS-936558 to the Physician's Choice of Either Dacarbazine or Carboplatin and Paclitaxel in Advanced Melanoma Patients That Have Progressed Following Anti-CTLA-4 Therapy (CheckMate 037)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-037; 2012-001828-35 (EudraCT Number)
Record Dates: First submitted 2012-11-02; First posted 2012-11-06 (Estimated); Results first posted 2017-03-22 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-03

CONDITIONS: Unresectable or Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; Dacarbazine; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BMS-936558 3 mg/kg (IV) (Experimental): BMS-936558 3 mg/kg solution for injection by intravenous (IV), every 2 weeks until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends
  Interventions: Biological: BMS-936558
- Investigator's Choice (Dacarbazine or Carboplatin+Paclitaxel) (Active Comparator): Dacarbazine: 1000mg/m2, Powder for IV solution, IV, every 3 weeks until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends
  Carboplatin: Area under the concentration-time curve (AUC) 6, solution for injection, IV, every 3 weeks until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends
  Paclitaxel: 175 mg/ m2, solution for injection, IV, every 3 weeks until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends
  Interventions: Drug: Dacarbazine; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Biological: BMS-936558
  Arms: BMS-936558 3 mg/kg (IV)
Drug: Dacarbazine
  Other Names: DTIC-Dome; DTIC
  Arms: Investigator's Choice (Dacarbazine or Carboplatin+Paclitaxel)
Drug: Carboplatin
  Other Names: Paraplatin; CBDCA
  Arms: Investigator's Choice (Dacarbazine or Carboplatin+Paclitaxel)
Drug: Paclitaxel
  Other Names: Onxol
  Arms: Investigator's Choice (Dacarbazine or Carboplatin+Paclitaxel)

SUMMARY:
The purpose of the study is to estimate the response rate and compare overall survival of patients taking BMS-936558 to those taking study physician's choice of either Dacarbazine or Carboplatin and Paclitaxel

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Men & women ≥ 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1
* Histologically confirmed Stage III (unresectable)/Stage IV melanoma
* Measurable disease by computed tomography (CT)/magnetic resonance imaging (MRI) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
* Objective evidence of disease progression (clinical or radiological) during or after at least 1 (V600 Wildtype) or at least 2 (V600 mutation positive) prior treatment regimens
* Pre-treatment fresh core, excision or punch tumor biopsy
* Archival Formalin-fixed paraffin-embedded (FFPE) tumor material if available

Exclusion Criteria:

* Any treatment in a BMS-936558 (Nivolumab) trial
* Subjects with condition requiring systemic treatment with either corticosteroids (> 10mg daily prednisone/equivalent) or other immunosuppressive medications within 14 days of study drug administration
* Active, known or suspected autoimmune disease
* Unknown BRAF status
* Active brain metastasis or leptomeningeal metastasis
* Ocular melanoma
* Prior therapy with anti programmed death-1 (anti-PD-1), anti programmed death-ligand 1 (anti-PD-L1) or anti-programmed death-ligand 2 (anti-PD-L2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2012-12-21 (Actual); Primary Completion 2016-02-16 (Actual); Study Completion 2020-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (91):
- United States (32):
  - Mayo Clinic, Phoenix, Arizona
  - UCSD Moores Cancer Center, La Jolla, California
  - The Angeles Clinic & Research Institute, Los Angeles, California
  - University Of California - Los Angeles, Los Angeles, California
  - San Francisco Oncology Associates, San Francciso, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - University Of Colorado, Aurora, Colorado
  - Yale University School Of Medicine, New Haven, Connecticut
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Orlando Health, Inc, Orlando, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Winship Cancer Institute, Atlanta, Georgia
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University Of Michigan Health System, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Allina Health, Minneapolis, Minnesota
  - Washington University School Of Medicine, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Clinical Cancer Center, New York, New York
  - MSKCC Clinical Laboratory at Nassau, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals, Cleveland, Ohio
  - Providence Oncology And Hematology, Portland, Oregon
  - Network Office of Research and Innovation, Allentown, Pennsylvania
  - St. Luke'S Health System, Allentown, Pennsylvania
  - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Huntsman Cancer Institute, Salt Lake City, Utah
- Austria (2):
  - Local Institution, Innsbruck
  - Local Institution, Vienna
- Belgium (3):
  - Local Institution, Brussels
  - Local Institution, Edegem
  - Local Institution, Leuven
- Brazil (3):
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Rio de Janeiro
  - Local Institution, São Paulo
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - Princess Margaret Hospital, Toronto, Ontario
  - CHUM, Montreal, Quebec
  - Sir Mortimer B Davis - Jewish General Hospital, Montreal, Quebec
- Denmark (3):
  - Aarhus Universitetshospital, Aarhus
  - Herlev Hospital, Herlev
  - Odense University Hospital, Odense
- France (8):
  - Local Institution, Clermont-Ferrand
  - Local Institution, Lille
  - Hopital La Timone, Marseille
  - Local Institution, Nantes
  - Local Institution, Nice
  - Local Institution, Paris
  - Local Institution, Pierre-Bénite
  - Local Institution, Villejuif
- Germany (12):
  - Local Institution, Würzburg, Bavaria
  - Local Institution, Buxtehude
  - Local Institution, Dresden
  - Local Institution, Essen
  - Local Institution, Frankfurt am Main
  - Local Institution, Hanover
  - Local Institution, Heidelberg
  - Local Institution, Kiel
  - Local Institution, Lübeck
  - Local Institution, Magdeburg
  - Local Institution, Munich
  - Local Institution, Tübingen
- Israel (2):
  - Local Institution, Jerusalem
  - Local Institution, Ramat Gan
- Italy (8):
  - Local Institution, Bari
  - Local Institution, Bergamo
  - Local Institution, Genova
  - Local Institution, Milan
  - Local Institution, Napoli
  - Local Institution, Padua
  - Local Institution, Roma
  - Local Institution, Siena
- Netherlands (3):
  - Local Institution, Amsterdam
  - Local Institution, Groningen
  - Local Institution, Maastricht
- Spain (4):
  - Local Institution, Barcelona
  - Local Institution, Madrid
  - Local Institution, Pamplona
  - Local Institution, Valencia
- Switzerland (2):
  - Local Institution, Lausanne
  - Local Institution, Zurich
- United Kingdom (5):
  - Local Institution, Manchester, Greater Manchester
  - Local Institution, Southampton, Hampshire
  - Local Institution, Oxford, Oxfordshire
  - Local Institution, Newcastle upon Tyne, Tyne and Wear
  - Local Institution, London

REFERENCES:
- [Derived] Larkin J, Minor D, D'Angelo S, Neyns B, Smylie M, Miller WH Jr, Gutzmer R, Linette G, Chmielowski B, Lao CD, Lorigan P, Grossmann K, Hassel JC, Sznol M, Daud A, Sosman J, Khushalani N, Schadendorf D, Hoeller C, Walker D, Kong G, Horak C, Weber J. Overall Survival in Patients With Advanced Melanoma Who Received Nivolumab Versus Investigator's Choice Chemotherapy in CheckMate 037: A Randomized, Controlled, Open-Label Phase III Trial. J Clin Oncol. 2018 Feb 1;36(4):383-390. doi: 10.1200/JCO.2016.71.8023. Epub 2017 Jul 3. PMID 28671856
- [Derived] Weber JS, D'Angelo SP, Minor D, Hodi FS, Gutzmer R, Neyns B, Hoeller C, Khushalani NI, Miller WH Jr, Lao CD, Linette GP, Thomas L, Lorigan P, Grossmann KF, Hassel JC, Maio M, Sznol M, Ascierto PA, Mohr P, Chmielowski B, Bryce A, Svane IM, Grob JJ, Krackhardt AM, Horak C, Lambert A, Yang AS, Larkin J. Nivolumab versus chemotherapy in patients with advanced melanoma who progressed after anti-CTLA-4 treatment (CheckMate 037): a randomised, controlled, open-label, phase 3 trial. Lancet Oncol. 2015 Apr;16(4):375-84. doi: 10.1016/S1470-2045(15)70076-8. Epub 2015 Mar 18. PMID 25795410
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 405 participants randomized and 370 treated.
Groups:
- Nivolumab: Nivolumab 3 mg/kg IV over 60 minutes Q2W
- Investigator's Choice (Dacarbazine or Carboplatin+Paclitaxel): Dacarbazine: 1000 mg/m^2 IV over 30 to 60 minutes Q3W, or Carboplatin: Area under the concentration-time curve (AUC) 6 IV over 30 minutes Q3W, and Paclitaxel: 175 mg/m^2 IV over 180 minutes Q3W
Period: Pre-Treatment
Arm/Group | Nivolumab | Investigator's Choice (Dacarbazine or Carboplatin+Paclitaxel)
Started (Started = Randomized) | 272 | 133
Completed (Completed = Received Treatment) | 268 | 102
Not Completed | 4 | 31
Not completed — Participant request to discontinue Study treatment | 0 | 13
Not completed — Withdrawal by Subject | 1 | 16
Not completed — Poor/Non-compliance | 1 | 0
Not completed — Participant no longer met study criteria | 2 | 2
Period: Treatment
Arm/Group | Nivolumab | Investigator's Choice (Dacarbazine or Carboplatin+Paclitaxel)
Started (Started = Received treatment) | 268 | 102
Completed (Completed = Completed treatment) | 0 | 0
Not Completed | 268 | 102
Not completed — Disease Progression | 192 | 74
Not completed — Study Drug Toxicity | 19 | 11
Not completed — Adverse Event unrelated to Study Drug | 6 | 3
Not completed — Participant request to discontinue Study treatment | 26 | 7
Not completed — Participant withdrew consent | 4 | 2
Not completed — Maximum Clinical Benefit | 9 | 3
Not completed — Poor/Non-compliance | 2 | 0
Not completed — Participant no longer met Study criteria | 4 | 0
Not completed — Other reasons | 6 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab | Investigator's Choice (Dacarbazine or Carboplatin+Paclitaxel) | Total
Number analyzed (Participants) | 272 | 133 | 405
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (14.1) | 60.3 (12.4) | 59.2 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 48 | 144
  Male | 176 | 85 | 261
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 116 | 61 | 177
  Unknown or Not Reported | 152 | 71 | 223
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 269 | 129 | 398
  Black or African American | 1 | 2 | 3
  Asian | 2 | 0 | 2
  American Indian or Alaska Native | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Objective response rate (ORR) per Independent Review Committee (IRC) is defined as the number of participants with a best overall response (BOR) of complete response (CR) or partial response (PR) divided by the number of randomized participants using RECIST 1.1
Time Frame: From date of randomization to the date of objectively documented progression, date of death, or the date of subsequent therapy (Up to approximately 38 months)
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab | Investigator's Choice (Dacarbazine or Carboplatin+Paclitaxel)
Number analyzed (Participants) | 272 | 133
Percentage of participants | 27.2 [22.0 to 32.9] | 9.8 [5.3 to 16.1]

2. Primary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) was defined the time between the date of randomization to the date of death. For participants without documentation of death, OS was censored on the last date the participant was known to be alive. Unit of measure (months) is the median survival time.
Time Frame: Up to 96 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Investigator's Choice (Dacarbazine or Carboplatin+Paclitaxel): Dacarbazine: 1000 mg/m^2 IV Q3W Carboplatin: Area under the concentration-time curve (AUC) 6 IV Q3W Paclitaxel: 175 mg/m^2 IV Q3W
Arm/Group | Nivolumab | Investigator's Choice (Dacarbazine or Carboplatin+Paclitaxel)
Number analyzed (Participants) | 272 | 133
Months | 15.74 [12.88 to 19.88] | 14.39 [11.66 to 18.17]
Statistical Analysis 1: Comparison: Nivolumab vs Investigator's Choice (Dacarbazine or Carboplatin+Paclitaxel); Hazard Ratio is Nivolumab 3 mg/kg (IV) over Investigator's Choice (Dacarbazine or Carboplatin+Paclitaxel); Test type: Superiority; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.68 to 1.08] — From stratified cox proportional hazard model with treatment group as a single covariate, stratified by BRAF status, prior anti-CTLA-4 benefit, and PD-L1 status (IVRS source)

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression Free Survival (PFS) is defined as the time from randomization to the date of the first documented progression, as determined by the Independent Review Committee (IRC) using RECIST 1.1, or death due to any cause, whichever occurs first. Participants who died without a reported progression were considered to have progressed on the date of their death. Participants who did not progress or die were censored on the date of their last evaluable tumor assessment before subsequent anti-cancer therapy. Unit of measure (months) is the median survival time.
Time Frame: From the date of randomization to the date of the first documented progression or death (Up to approximately 38 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab | Investigator's Choice (Dacarbazine or Carboplatin+Paclitaxel)
Number analyzed (Participants) | 272 | 133
months | 3.12 [2.33 to 3.52] | 3.65 [2.30 to 5.29]
Statistical Analysis 1: Comparison: Nivolumab vs Investigator's Choice (Dacarbazine or Carboplatin+Paclitaxel); Hazard Ratio is Nivolumab 3 mg/kg (IV) over Investigator's Choice (Dacarbazine or Carboplatin+Paclitaxel); Test type: Superiority; Hazard Ratio (HR) = 1.03, 95.1% CI 2-sided [0.78 to 1.36] — Stratified Cox proportional hazard model

4. Secondary Outcome: Objective Response Rate (ORR) by Baseline PD-L1 Expression
Description: Objective Response Rate (ORR) is defined as the number of participants with a Best Overall Response (BOR) of complete response (CR) or partial response (PR) divided by number of randomized participants. PD-L1 expression evaluated for ORR.
Time Frame: From date of randomization to the date of objectively documented progression or the date of subsequent therapy (Up to approximately 38 months)
Population: All PD-L1 Evaluable Participants for ORR
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab | Investigator's Choice (Dacarbazine or Carboplatin+Paclitaxel)
Number analyzed (Participants) | 267 | 131
Percentage of participants
  <5% PD-L1 expression: number analyzed (Participants) | 137 | 58
  <5% PD-L1 expression | 15.3 [9.7 to 22.5] | 13.8 [6.1 to 25.4]
  >=5% PD-L1 expression: number analyzed (Participants) | 111 | 41
  >=5% PD-L1 expression | 43.2 [33.9 to 53.0] | 12.2 [4.1 to 26.2]
Statistical Analysis 1: Comparison: Nivolumab vs Investigator's Choice (Dacarbazine or Carboplatin+Paclitaxel); For <5% PD-L1 expression. Ratio of Nivolumab over Investigator's Choice; Test type: Superiority; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.44 to 3.16]
Statistical Analysis 2: Comparison: Nivolumab vs Investigator's Choice (Dacarbazine or Carboplatin+Paclitaxel); For >=5% PD-L1 expression. Ratio of Nivolumab over Investigator's Choice; Test type: Superiority; Odds Ratio (OR) = 5.49, 95% CI 2-sided [1.92 to 19.08]

5. Secondary Outcome: Overall Survival (OS) by PD-L1 Positive
Description: Overall Survival (OS) by PD-L1 expression was defined the time between the date of randomization to the date of death. For participants without documentation of death, OS was censored on the last date the participant was known to be alive.
Time Frame: Up to 96 months
Population: All PD-L1 positive evaluable participants for OS
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab | Investigator's Choice (Dacarbazine or Carboplatin+Paclitaxel)
Number analyzed (Participants) | 135 | 67
Months | 31.44 [20.57 to 46.69] | 16.72 [11.83 to 31.44]
Statistical Analysis 1: Comparison: Nivolumab vs Investigator's Choice (Dacarbazine or Carboplatin+Paclitaxel); PD-L1 Positive; Test type: Superiority; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.50 to 1.01] — From unstratified Cox proportional hazard model

6. Secondary Outcome: Overall Survival (OS) by PD-L1 Negative
Description: as for outcome 5
Time Frame: Up to 96 months
Population: All PD-L1 negative evaluable participants for OS
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab | Investigator's Choice (Dacarbazine or Carboplatin+Paclitaxel)
Number analyzed (Participants) | 137 | 66
Months | 11.14 [7.72 to 13.21] | 11.76 [8.05 to 17.81]
Statistical Analysis 1: Comparison: Nivolumab vs Investigator's Choice (Dacarbazine or Carboplatin+Paclitaxel); PD-L1 Negative; Test type: Superiority; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.75 to 1.41] — From unstratified Cox proportional hazard model

7. Secondary Outcome: Mean Change From Baseline in Health-related Quality of Life (HRQoL)
Description: Health-related Quality of Life (HRQoL) was assessed with the EORTC QLQ-C30 questionnaire, which is the most commonly used quality-of-life instrument in oncology trials. The instrument's 30 items were divided among 5 functional scales (physical, role, cognitive, emotional, and social), 9 symptom scales (fatigue, pain, nausea/vomiting, dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties), and a global health/quality of life scale. Raw scores for the EORTC QLQ-C30 were transformed to a 0-100 metric.
  Higher scores for all functional scales and Global Health Status=better HRQoL Increase from baseline indicates improvement in HRQoL. Lower scores for symptom scales=better HRQoL Decline from baseline for symptom scales =improvement in symptoms compared to baseline.
  A 10 point difference on a 100 point scale between treatments was considered clinically significant.
Time Frame: From Baseline (Day1) to second Follow-Up (Up to 96 months)
Population: All randomized participants
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Nivolumab | Investigator's Choice (Dacarbazine or Carboplatin+Paclitaxel)
Number analyzed (Participants) | 272 | 133
Units on a scale
  Physical Functioning Follow-Up 1: number analyzed (Participants) | 77 | 22
  Physical Functioning Follow-Up 1 | -7.97 (20.49) | -12.73 (21.47)
  Physical Functioning Follow-Up 2: number analyzed (Participants) | 62 | 28
  Physical Functioning Follow-Up 2 | -3.66 (16.05) | -7.14 (16.02)
  Role Functioning Follow-Up 1: number analyzed (Participants) | 77 | 22
  Role Functioning Follow-Up 1 | -14.94 (31.13) | -15.91 (29.76)
  Role Functioning Follow-Up 2: number analyzed (Participants) | 62 | 28
  Role Functioning Follow-Up 2 | -7.80 (25.56) | -8.33 (21.52)
  Emotional Functioning Follow-Up 1: number analyzed (Participants) | 77 | 21
  Emotional Functioning Follow-Up 1 | -5.09 (21.59) | -15.48 (24.48)
  Emotional Functioning Follow-Up 2: number analyzed (Participants) | 62 | 28
  Emotional Functioning Follow-Up 2 | -0.94 (19.15) | -5.36 (25.98)
  Cognitive Functioning Follow-Up 1: number analyzed (Participants) | 77 | 21
  Cognitive Functioning Follow-Up 1 | -7.58 (16.79) | -7.94 (17.17)
  Cognitive Functioning Follow-Up 2: number analyzed (Participants) | 62 | 28
  Cognitive Functioning Follow-Up 2 | -3.49 (15.43) | -1.19 (13.55)
  Social Functioning Follow-Up 1: number analyzed (Participants) | 77 | 21
  Social Functioning Follow-Up 1 | -8.66 (29.45) | -18.25 (26.82)
  Social Functioning Follow-Up 2: number analyzed (Participants) | 62 | 28
  Social Functioning Follow-Up 2 | -1.61 (29.52) | -4.17 (24.69)
  Global Health Status Follow-Up 1: number analyzed (Participants) | 77 | 21
  Global Health Status Follow-Up 1 | -8.23 (22.44) | -10.71 (17.71)
  Global Health Status Follow-Up 2: number analyzed (Participants) | 62 | 28
  Global Health Status Follow-Up 2 | -1.61 (18.53) | -3.27 (12.07)
  Dyspnea Follow-Up 1: number analyzed (Participants) | 77 | 22
  Dyspnea Follow-Up 1 | 6.06 (27.96) | 16.67 (24.67)
  Dyspnea Follow-Up 2: number analyzed (Participants) | 62 | 28
  Dyspnea Follow-Up 2 | 5.91 (22.20) | 7.14 (24.61)
  Insomnia Follow-Up 1: number analyzed (Participants) | 77 | 22
  Insomnia Follow-Up 1 | 3.46 (32.26) | 0.00 (30.86)
  Insomnia Follow-Up 2: number analyzed (Participants) | 62 | 28
  Insomnia Follow-Up 2 | -4.84 (25.50) | 0.00 (30.09)
  Apatite loss Follow-Up 1: number analyzed (Participants) | 77 | 22
  Apatite loss Follow-Up 1 | 6.93 (28.79) | 13.64 (24.47)
  Apatite loss Follow-Up 2: number analyzed (Participants) | 62 | 28
  Apatite loss Follow-Up 2 | 5.91 (30.49) | 2.38 (22.09)
  Constipation Follow-Up 1: number analyzed (Participants) | 77 | 21
  Constipation Follow-Up 1 | 7.36 (28.93) | 0.00 (23.57)
  Constipation Follow-Up 2: number analyzed (Participants) | 62 | 28
  Constipation Follow-Up 2 | 2.15 (22.48) | -2.38 (29.99)
  Diarrhea Follow-Up 1: number analyzed (Participants) | 77 | 21
  Diarrhea Follow-Up 1 | -0.43 (19.86) | 6.35 (22.65)
  Diarrhea Follow-Up 2: number analyzed (Participants) | 62 | 28
  Diarrhea Follow-Up 2 | 1.08 (20.88) | 1.19 (16.93)
  Financial Difficulties Follow-Up 1: number analyzed (Participants) | 77 | 21
  Financial Difficulties Follow-Up 1 | -1.73 (25.87) | 4.76 (39.84)
  Financial Difficulties Follow-Up 2: number analyzed (Participants) | 62 | 28
  Financial Difficulties Follow-Up 2 | -1.08 (22.56) | -2.38 (28.59)
  Fatigue Follow-Up 1: number analyzed (Participants) | 77 | 22
  Fatigue Follow-Up 1 | 8.95 (23.78) | 15.66 (28.00)
  Fatigue Follow-Up 2: number analyzed (Participants) | 62 | 28
  Fatigue Follow-Up 2 | 4.84 (22.55) | 7.14 (21.85)
  Nausea and Vomiting Follow-Up 1: number analyzed (Participants) | 77 | 22
  Nausea and Vomiting Follow-Up 1 | 2.81 (17.19) | 10.61 (25.48)
  Nausea and Vomiting Follow-Up 2 | 0.00 (15.39) | 2.98 (18.73)
  Pain Follow-Up 1: number analyzed (Participants) | 77 | 22
  Pain Follow-Up 1 | 6.06 (31.17) | 6.82 (25.02)
  Pain Follow-Up 2 | 5.38 (24.84) | -1.79 (14.59)

ADVERSE EVENTS:
Time Frame: From first dose to 100 days post last dose (Up to 96 months)
Arm/Group | Nivolumab | Investigator's Choice (Dacarbazine or Carboplatin+Paclitaxel)
All-Cause Mortality (participants affected / at risk) | 206/268 | 88/102
Serious Adverse Events (participants affected / at risk) | 191/268 | 37/102
Other Adverse Events (participants affected / at risk) | 255/268 | 95/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab (N=268) | Investigator's Choice (Dacarbazine or Carboplatin+Paclitaxel) (N=102)
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Blood loss anaemia (Blood and lymphatic system disorders) | 1 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0
Splenic haematoma (Blood and lymphatic system disorders) | 1 | 0
Splenic lesion (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 0
Atrial flutter (Cardiac disorders) | 2 | 0
Cardiac arrest (Cardiac disorders) | 3 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 2 | 0
Adrenal haemorrhage (Endocrine disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 2 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 2
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Intestinal fistula (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 1
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 3 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 3
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Fatigue (General disorders) | 2 | 2
Gait disturbance (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 6 | 0
Infusion site extravasation (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Pain (General disorders) | 1 | 2
Pelvic mass (General disorders) | 1 | 0
Pyrexia (General disorders) | 5 | 2
Ulcer (General disorders) | 1 | 0
Biliary obstruction (Hepatobiliary disorders) | 1 | 0
Hepatic haemorrhage (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 2 | 0
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Bronchitis bacterial (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 2 | 1
Febrile infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 8 | 0
Pneumonia pseudomonal (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 4 | 0
Urinary tract infection (Infections and infestations) | 3 | 0
Urosepsis (Infections and infestations) | 1 | 0
Vascular device infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 2 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Open fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0
Radiation necrosis (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 1
Vascular access site thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Ejection fraction abnormal (Investigations) | 1 | 0
General physical condition abnormal (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Influenza B virus test positive (Investigations) | 1 | 0
Lipase increased (Investigations) | 2 | 0
Liver function test abnormal (Investigations) | 1 | 0
Liver function test increased (Investigations) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 86 | 18
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Skin neoplasm bleeding (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour fistulisation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Aphasia (Nervous system disorders) | 1 | 0
Autoimmune neuropathy (Nervous system disorders) | 1 | 0
Brain oedema (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 1
Demyelination (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Facial paresis (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 3 | 0
Headache (Nervous system disorders) | 1 | 0
Incoherent (Nervous system disorders) | 0 | 1
Monoplegia (Nervous system disorders) | 1 | 0
Paraplegia (Nervous system disorders) | 1 | 0
Post herpetic neuralgia (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 2 | 0
Status epilepticus (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
VIth nerve paralysis (Nervous system disorders) | 1 | 0
Burnout syndrome (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 3 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 2
Hydronephrosis (Renal and urinary disorders) | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 2 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Embolism (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 3 | 1
Peripheral embolism (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab (N=268) | Investigator's Choice (Dacarbazine or Carboplatin+Paclitaxel) (N=102)
Anaemia (Blood and lymphatic system disorders) | 65 | 31
Leukopenia (Blood and lymphatic system disorders) | 4 | 10
Neutropenia (Blood and lymphatic system disorders) | 3 | 24
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 11
Hypothyroidism (Endocrine disorders) | 27 | 0
Abdominal pain (Gastrointestinal disorders) | 50 | 13
Abdominal pain upper (Gastrointestinal disorders) | 21 | 6
Constipation (Gastrointestinal disorders) | 53 | 23
Diarrhoea (Gastrointestinal disorders) | 90 | 18
Dry mouth (Gastrointestinal disorders) | 14 | 3
Dyspepsia (Gastrointestinal disorders) | 21 | 4
Nausea (Gastrointestinal disorders) | 91 | 43
Vomiting (Gastrointestinal disorders) | 57 | 24
Asthenia (General disorders) | 35 | 11
Chills (General disorders) | 18 | 3
Fatigue (General disorders) | 135 | 52
Influenza like illness (General disorders) | 20 | 4
Oedema peripheral (General disorders) | 44 | 5
Pain (General disorders) | 27 | 4
Pyrexia (General disorders) | 52 | 10
Nasopharyngitis (Infections and infestations) | 26 | 4
Upper respiratory tract infection (Infections and infestations) | 25 | 2
Urinary tract infection (Infections and infestations) | 24 | 4
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 9
Alanine aminotransferase increased (Investigations) | 29 | 4
Aspartate aminotransferase increased (Investigations) | 38 | 6
Blood alkaline phosphatase increased (Investigations) | 22 | 3
Blood creatinine increased (Investigations) | 20 | 2
Neutrophil count decreased (Investigations) | 1 | 8
Platelet count decreased (Investigations) | 11 | 9
Weight decreased (Investigations) | 25 | 8
White blood cell count decreased (Investigations) | 7 | 9
Decreased appetite (Metabolism and nutrition disorders) | 54 | 21
Hyperglycaemia (Metabolism and nutrition disorders) | 14 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 14 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 20 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 15 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 15 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 25 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 76 | 21
Back pain (Musculoskeletal and connective tissue disorders) | 55 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 16 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 31 | 10
Neck pain (Musculoskeletal and connective tissue disorders) | 15 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 37 | 13
Dizziness (Nervous system disorders) | 30 | 5
Headache (Nervous system disorders) | 47 | 11
Neuropathy peripheral (Nervous system disorders) | 10 | 11
Paraesthesia (Nervous system disorders) | 13 | 13
Anxiety (Psychiatric disorders) | 19 | 1
Depression (Psychiatric disorders) | 8 | 6
Insomnia (Psychiatric disorders) | 34 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 73 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 52 | 14
Alopecia (Skin and subcutaneous tissue disorders) | 8 | 30
Dry skin (Skin and subcutaneous tissue disorders) | 24 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 73 | 2
Rash (Skin and subcutaneous tissue disorders) | 57 | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 22 | 2
Vitiligo (Skin and subcutaneous tissue disorders) | 31 | 1
Hypertension (Vascular disorders) | 21 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.